CLINICAL TRIAL: NCT02504918
Title: Markers of T Cell Suppression: Associations With Malaria Infection and Antimalarial Treatment
Brief Title: Markers of T Cell Suppression: Associations With Malaria Infection and Antimalarial Treatment in Malian Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915163; 15-I-N163
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06-12

CONDITIONS: Malaria
Keywords: Plasmodium Falciparum; Regulatory; Chemoprevention; Coartem; Parasitemia
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Parasitemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- The disease malaria can cause very serious health problems. Researchers want to see if malaria affects the way T cells and vaccines work in the body. If it does, they may need to give malaria treatments before vaccines. They want to check the T cells in children who do or do not get antimalarial treatment.

Objectives:

- To study the effect of blood stage malaria on T cell suppression and vaccine responses. To describe markers of T cell suppression in children who do or do not receive antimalarial treatment.

Eligibility:

- Children ages 12 59 months living near Ouelessebougou in Mali. They must have no serious illness.

Design:

* Participants will be screened with medical history and physical exam.
* Some participants will get a course of antimalarial tablets. Some will not. This will be decided at random.
* Participants will have monthly visits for up to a year. They will have blood tests at each visit.

DETAILED DESCRIPTION:
Malaria caused by Plasmodium falciparum continues to be a global problem with devastating consequences. New interventions are needed to combat malaria, and progress is being made in development of vaccines: a subunit vaccine called RTSS confers partial protection against clinical malaria in children and is nearing licensure; a whole organism product called PfSPZ Vaccine can confer sterile protection against infection, and is now undergoing field trials. NIAID is involved in field trials of PfSPZ Vaccine and other vaccines, and a key question in vaccine trial design has been whether concurrent parasitemia will impair vaccine responses. The primary hypothesis in this study is that T cell suppression and regulation will decrease following antimalarial treatment that clears blood stage parasites for an extended period of time.

Up to 200 children will be recruited into longitudinal studies that will be conducted in Ouelessebougou and neighboring villages in Mali. In August 2015, up to 50 children presenting for Seasonal Malaria Chemoprevention (SMC) in a village where the government has implemented SMC will be enrolled, as well as up to 50 age-matched children residing in an adjacent village where SMC has not been implemented by the government of Mali; and then followed through the rainy season. In January 2016, up to 100 healthy children in Ouelessebougou village area will be enrolled and randomized to receive or not receive a course of artemether-lumefantrine, and then followed for the duration of the dry season (Jan-Jun 2016) and the subsequent rainy season (Jul-Dec 2016). Samples in both cohort studies (age-matched SMC study; randomized artemether-lumefantrine study) will be collected from the children at the time of monthly visits and assessed in ex vivo assays for markers of T cell suppression as the primary outcome of this study. For our secondary outcomes, we will examine levels of regulatory T cells, measure T cell responses in stimulation assays, and survey parasitemia by blood smear and by polymerase chain reaction (PCR) assays. We expect that levels of T cell suppression and regulatory T cells will be similar between groups before antimalarial treatment or malaria infection, but after treatment or in those subjects that remain uninfected these levels will be significantly lower as compared to the untreated and or infected subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

A study participant must satisfy the following criteria to be enrolled in this study:

* A child between 12-59 months
* Parent/guardian able to provide consent
* Resident of the health district of Ouelessebougou or neighboring district for at least a year

EXCLUSION CRITERIA:

* Clinically symptomatic or apparent severe anemia or any other condition that may be worsened by 5 mL phlebotomy or any other study procedure
* Chronic or debilitating condition that precludes attendance for monthly visits
* Known or clinically apparent condition of immunosuppression or chronic infection.
* Known allergies to study treatments (SP; amodiaquine; artemether-lumefantrine)
* Use of cotrimaxozale on a routine basis for prophylaxis
* Conditions that in the judgment of the investigator could increase the risk to the volunteer.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-07-21; Primary Completion 2016-12-31 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
To investigate the association of recent malaria infection and percentage of PD1+ CD4 T cells in children that have not received SMC during the rainy season. | Approximately 3-6 months
To compare the percentage of PD1 +CD4 T cells in children who do or do not receive antimalarial treatment, in both rainy season and drythedry season. | Approximately 3-6 months

SECONDARY OUTCOMES:
To compare and describe levels of regulatory T cells in children who do or do not receive antimalarial treatment, in both rainy season and dry season. To compare and describe T cell stimulation responses in children who do or do not receive anti... | Approximately 3-6 months
To determine and investigate phenotypic differences in T cell subsets in infected and uninfected subjects at baseline. | Approximately 3-6 months
To confirm that blood stage parasite burden is markedly reduced throughout the dry season by a single treatment with artemether-lumefantrine at enrollment; and to examine the association of parasite clearance during the dry season on malaria ris... | Approximately 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fried, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ouelessebougou Clinical Research Center MRTC/ FMPOS, Wolossébougou, Mali

REFERENCES:
- [Background] Cunnington AJ, Riley EM. Suppression of vaccine responses by malaria: insignificant or overlooked? Expert Rev Vaccines. 2010 Apr;9(4):409-29. doi: 10.1586/erv.10.16. PMID 20370551
- [Background] Dicko A, Diallo AI, Tembine I, Dicko Y, Dara N, Sidibe Y, Santara G, Diawara H, Conare T, Djimde A, Chandramohan D, Cousens S, Milligan PJ, Diallo DA, Doumbo OK, Greenwood B. Intermittent preventive treatment of malaria provides substantial protection against malaria in children already protected by an insecticide-treated bednet in Mali: a randomised, double-blind, placebo-controlled trial. PLoS Med. 2011 Feb 1;8(2):e1000407. doi: 10.1371/journal.pmed.1000407. PMID 21304923
- [Background] Wilson AL; IPTc Taskforce. A systematic review and meta-analysis of the efficacy and safety of intermittent preventive treatment of malaria in children (IPTc). PLoS One. 2011 Feb 14;6(2):e16976. doi: 10.1371/journal.pone.0016976. PMID 21340029
- [Derived] Attaher O, Zaidi I, Kwan JL, Issiaka D, Samassekou MB, Cisse KB, Coulibaly B, Keita S, Sissoko S, Traore T, Diarra K, Diarra BS, Dembele A, Kanoute MB, Mahamar A, Barry A, Fried M, Dicko A, Duffy PE. Effect of Seasonal Malaria Chemoprevention on Immune Markers of Exhaustion and Regulation. J Infect Dis. 2020 Jan 1;221(1):138-145. doi: 10.1093/infdis/jiz415. PMID 31584094